CLINICAL TRIAL: NCT02362035
Title: A Phase 1b/2 Proof-of-Concept Study of the Combination of ACP-196 (Acalabrutinib) and Pembrolizumab in Subjects With Hematologic Malignancies
Brief Title: ACP-196 (Acalabrutinib) in Combination With Pembrolizumab, for Treatment of Hematologic Malignancies
Acronym: KEYNOTE145
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-LY-005
Record Dates: First submitted 2015-02-07; First posted 2015-02-12 (Estimated); Results first posted 2022-05-06 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Follicular Lymphoma (FL); CLL; Small Lymphocytic Lymphoma (SLL); Richter's Syndrome; Mantle Cell Lymphoma (MCL); Indolent Non Hodgkin Lymphoma; Waldenström Macroglobulinemia; Multiple Myeloma; Hodgkin Lymphoma; Burkitt Lymphoma; Marginal Zone Lymphomas; Mediastinal Large B Cell Lymphoma; Hairy Cell Leukemia
Keywords: Bruton tyrosine kinase inhibitor; Btk; B-Cell Malignancies; Mantle Cell; Multiple Myeloma; CLL; SLL; DLBCL; Follicular; Waldenstrom; Burkitt lymphoma; marginal zone lymphomas; hairy cell leukemia; B cell acute lymphoid leukemia; Acalabrutinib; ACP-196
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Multiple Myeloma; Hodgkin Disease; Burkitt Lymphoma; Leukemia, Hairy Cell | interventions — acalabrutinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acalabrutinib plus Pembrolizumab (Experimental): A nonrandomized study that will be conducted in 2 stages. In the first stage, (Safety), subjects will receive Acalabrutinib Dose A orally administered (PO) twice daily (BID) in combination with Pembrolizumab Dose B administered every 3 weeks (Q3W).
  The second stage was an expansion of Cohorts with the same dose regimen as the first stage. An additional expansion in subjects with Myelofibrosis was planned but not conducted.
  Interventions: Drug: Acalabrutinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Acalabrutinib — Orally Administered (PO)
  Other Names: ACP-196
Drug: Pembrolizumab — Intravenous Administered (IV)
  Other Names: KEYTRUDA

SUMMARY:
This study is evaluating the safety, pharmacodynamics (PD), and efficacy of acalabrutinib and pembrolizumab in hematologic malignancies.

DETAILED DESCRIPTION:
This is a Phase 1b/2, open-label, nonrandomized study that will be conducted in 2 stages. In the first stage, Part 1 of the study will determine the safety and preliminary efficacy of acalabrutinib and pembrolizumab in a limited group of B-cell malignancies. In the second stage, Part 2 allows for possible expansion cohorts into a wider range of B-cell malignancies, and Part 3 will evaluate the combination in subjects with myelofibrosis (MF).

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of a hematologic malignancy as documented by medical records and with histology based on criteria established by the World Health Organization (WHO).
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
* Agreement to use contraception during the study and for 90 days after the last dose of ACP-196 or 120 days after the last dose of pembrolizumab, if sexually active and able to bear or beget children.
* Completion of all therapy (including surgery, radiotherapy, chemotherapy, immunotherapy, or investigational therapy) for the treatment of cancer ≥ 4 weeks before the start of study therapy.
* ANC ≥ 0.5 x 10^9/L or platelet count ≥ 50 x 10^9/L unless due to disease involvement in the bone marrow.

Main Exclusion Criteria:

* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of study drugs, or put the study outcomes at undue risk.
* Central nervous system (CNS) involvement by lymphoma/leukemia
* Any therapeutic antibody within 4 weeks of first dose of study drugs.
* Total bilirubin > 1.5 x ULN; and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3.0 x ULN.
* Estimated creatinine clearance of < 30 mL/min, calculated using the formula of Cockcroft and Gault (140-Age) • Mass (kg)/(72 • creatinine mg/dL); multiply by 0.85 if female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2025-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Clinical Study Information Center, Study Director — 1-877-240-9479 - information.center@astrazeneca.com
Locations (19):
- United States (19):
  - Research Site, Tucson, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Denver, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Niles, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Columbus, Ohio
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Vancouver, Washington
  - Research Site, Yakima, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-005&attachmentIdentifier=2ded1a27-c5da-4fed-8db9-94e3d52b3efe&fileName=ACE-LY-005_RedactedCSP.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-005&attachmentIdentifier=1f7042f3-d331-4fc2-a94c-958b96d3518e&fileName=ACE-LY-005_RedactedSAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For the ACE-LY-005 program, Study Terminated by Sponsor refers to the following: Patients receiving treatment benefits will continue to be provided with study medication in the Post Final Analysis Management of the trial. No further data collection for analysis and reporting will be completed after the final Analysis
Groups:
- Acalabrutinib + Pembrolizumab: All participants in this study received both study drugs and were therefore analysed together as a single treatment arm.
  Participants receiving the different regimens were not analysed separately by regimen, as the study was designed to assess the safety of the combination study treatment.
  The study included N=161 participants who received both acalabrutinib and pembrolizumab and are summarized together (from First stage safety lead-in and Second stage expansion). Stage 3 (additional expansion in subjects with Myelofibrosis) was planned but not conducted.
Period: Overall Study
Arm/Group | Acalabrutinib + Pembrolizumab
Started | 161
Completed | 0
Not Completed | 161
Not completed — Death | 67
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Subject started another cancer therapy | 10
Not completed — Study terminated by sponsor | 45
Not completed — Decision by subject not related to AE/SAE | 2
Not completed — Decision by PI not related to AE/SAE | 1
Not completed — Disease progression | 11
Not completed — Withdrawal by Subject | 20

BASELINE CHARACTERISTICS:
Population: All participants in this study received both study drugs and were therefore analyzed together as a single treatment arm. Participants receiving the different regimens were not analyzed separately by regimen, as the study was designed to assess the safety of the combination study treatment.
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 98
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 148
  Not Reported | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Black or African American | 5
  Native Hawaiian or Other Pacific Islander | 2
  White | 141
  Not Reported | 9
Region of Enrollment [Number; unit: Participants]
  USA | 161

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: Treatment-emergent AEs were defined as those events that occurred on or after the first dose of study drug, through the treatment phase, and within 30 days following the last dose of study drug.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 160

2. Primary Outcome: Number of Participants With Grade 3-4 Adverse Events
Description: Severity of AEs was graded using the Common Terminology Criteria for Adverse Events (CTCAE), version 4.03
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 105

3. Primary Outcome: Number of Participants With Grade 5 Adverse Events
Description: Number of participants with CTCAE Grade 5 (fatal) adverse events
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 9

4. Primary Outcome: Number of Participants With Any Study-Drug Related AE
Description: Study drug-related AEs were those assessed by investigator as related to study treatment.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 142

5. Primary Outcome: Number of Participants With Grade 3-4 Study-Drug Related AE
Description: The severity of the AEs was assessed by NCI CTCAE Version 4.03 or higher. Drug-related AEs were those assessed by investigator as related to study treatment.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 66

6. Primary Outcome: Number of Participants With Grade 5 Study-Drug Related AE
Description: Grade 5 (fatal) AEs assessed by investigator as related to study treatment.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 3

7. Primary Outcome: Number of Participants With Any SAE
Description: Serious AEs were those that resulted in death, were life-threatening, required or prolonged in-patient hospitalization, resulted in persistent or significant disability/incapacity, resulted in a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product, or were considered a significant medical event by the investigator based on medical judgment.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 75

8. Primary Outcome: Number of Participants With Grade 3-4 Any SAE
Description: Serious AEs were those that resulted in death, were life-threatening, required or prolonged in-patient hospitalization, resulted in persistent or significant disability/incapacity, resulted in a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product, or were considered a significant medical event by the investigator based on medical judgment. The severity of the AEs was assessed by NCI CTCAE Version 4.03 or higher.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 64

9. Primary Outcome: Number of Participants With Grade 5 Any SAE
Description: Grade 5 events were fatal events. Serious AEs were those that resulted in death, were life-threatening, required or prolonged in-patient hospitalization, resulted in persistent or significant disability/incapacity, resulted in a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product, or were considered a significant medical event by the investigator based on medical judgment.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 9

10. Primary Outcome: Number of Participants With Any Study Drug-Related SAE
Description: Serious AEs were those that resulted in death, were life-threatening, required or prolonged in-patient hospitalization, resulted in persistent or significant disability/incapacity, resulted in a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product, or were considered a significant medical event by the investigator based on medical judgment. Drug-related AEs were those assessed by investigator as related to study treatment.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 34

11. Primary Outcome: Number of Participants With Any Grade 3-4 Study Drug-Related SAE
Description: Serious AEs were those that resulted in death, were life-threatening, required or prolonged in-patient hospitalization, resulted in persistent or significant disability/incapacity, resulted in a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product, or were considered a significant medical event by the investigator based on medical judgment. The severity of the AEs was assessed by NCI CTCAE Version 4.03 or higher. Drug-related AEs were those assessed by investigator as related to study treatment.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 30

12. Primary Outcome: Number of Participants With Any Grade 5 Study Drug-Related SAE
Description: Grade 5 AEs were fatal events. Serious AEs were those that resulted in death, were life-threatening, required or prolonged in-patient hospitalization, resulted in persistent or significant disability/incapacity, resulted in a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product, or were considered a significant medical event by the investigator based on medical judgment. Drug-related AEs were those assessed by investigator as related to study treatment.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 3

13. Primary Outcome: Number of Participants With AE Leading to Study Drug Discontinuation, Modification or Delay
Description: AEs that discontinuation of study treatment, or a reduction in dosage, or a delay (temporary withholding) in treatment.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 83

14. Primary Outcome: Number of Participants With AE Leading to Study Drug Discontinuation
Description: An adverse event that resulted in the permanent discontinuation of study treatment in the study.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 45

15. Primary Outcome: Number of Participants With AE Leading to Study Drug Delay
Description: An adverse event that caused a temporary withholding of study treatment.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 71

16. Primary Outcome: Number of Participants With AE Leading to Study Drug Modification
Description: An adverse event that resulted in a reduction in the dosage of study treatment for that participant.
Time Frame: 104 weeks
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Number of participants | 9

17. Secondary Outcome: Overall Response Rate
Description: The percentage of subjects who achieve a partial response or complete response
Time Frame: 104 weeks
Population: All participants in this study received both study drugs and were therefore analyzed together as a single treatment arm. Participants receiving the different regimens were not analyzed separately by regimen, as the study was designed to assess the the combination study treatment.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
percent | 38.5 [31.0 to 46.5]

18. Secondary Outcome: Duration of Response
Description: The interval from the first documentation of response to the earlier of the first documentation of definitive disease progression or death from any cause
Time Frame: 104 weeks
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Months | 28.5 [9.0 to 36.4]

19. Secondary Outcome: Progression-free Survival
Description: The interval from the first dose date of acalabrutinib or pembrolizumab to the earlier of the first documentation of objective disease progression or death from any cause
Time Frame: 104 weeks
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Months | 4.7 [3.3 to 6.9]

20. Secondary Outcome: Overall Survival
Description: The time from the first dose date of acalabrutinib or pembrolizumab until date of death due to any cause
Time Frame: 104 weeks
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Months | 50.4 [26.2 to NA] — NA= not estimable. The NA of the 95% upper bound was calculated from the median. Since the upper limit of the KM curve hadn't reached 50%, there is no estimate for the upper confidence limit on the median. Therefore it's NA = not estimable.

21. Secondary Outcome: Time to Next Treatment
Description: The time from the first dose date of acalabrutinib or pembrolizumab to the start of the next treatment other than the study treatment
Time Frame: 104 weeks
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Acalabrutinib + Pembrolizumab
Number analyzed (Participants) | 161
Months | 21.1 [10.5 to 34.7]

ADVERSE EVENTS:
Time Frame: For each subject, adverse event data were collected from first dose of study drug until 30 days after the last dose, until the end of the study (data cutoff date of 14 July 2020).
Description: All participants in this study received both study drugs and were analyzed together as a single treatment arm. There were 3 Stages to the study (representing different disease histologies) and not 3 arms in the study. Study data are presented by disease histology for all subjects in Stage 1 (N=30) and Stage 2 (N=131) as TOTAL subjects (N=161). Stage 3 of the study was not conducted.
Arm/Group | Acalabrutinib + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 69/161
Serious Adverse Events (participants affected / at risk) | 75/161
Other Adverse Events (participants affected / at risk) | 157/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib + Pembrolizumab (N=161)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (3)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Retroperitoneal mass (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2)
Epiglottitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Meningitis bacterial (Infections and infestations) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 9 (9)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 5 (5)
Septic shock (Infections and infestations) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyponatraemic seizure (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (3)
Mental status changes (Psychiatric disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Renal failure (Renal and urinary disorders) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib + Pembrolizumab (N=161)
Anaemia (Blood and lymphatic system disorders) | 35 (56)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Lymph node pain (Blood and lymphatic system disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 16 (27)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (20)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (9)
Atrial flutter (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 2 (2)
Extrasystoles (Cardiac disorders) | 1 (1)
Myocardial calcification (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3)
Pericardial effusion (Cardiac disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (6)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (5)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (2)
Ear congestion (Ear and labyrinth disorders) | 3 (3)
Ear discomfort (Ear and labyrinth disorders) | 2 (2)
Ear haemorrhage (Ear and labyrinth disorders) | 2 (2)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Borderline glaucoma (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Chalazion (Eye disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 2 (2)
Eye pruritus (Eye disorders) | 1 (1)
Eyelid rash (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1)
Periorbital swelling (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 6 (6)
Vitreous degeneration (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 11 (17)
Abdominal pain (Gastrointestinal disorders) | 13 (18)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 10 (11)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (3)
Colitis microscopic (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 20 (21)
Diarrhoea (Gastrointestinal disorders) | 73 (135)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 8 (9)
Dysphagia (Gastrointestinal disorders) | 9 (9)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 4 (4)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Gingival discomfort (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Hyperaesthesia teeth (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 43 (63)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (3)
Palatal disorder (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (7)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 33 (45)
Asthenia (General disorders) | 12 (13)
Axillary pain (General disorders) | 2 (2)
Catheter site pain (General disorders) | 1 (1)
Chest discomfort (General disorders) | 2 (3)
Chills (General disorders) | 13 (16)
Drug withdrawal syndrome (General disorders) | 1 (1)
Early satiety (General disorders) | 1 (1)
Exercise tolerance decreased (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 57 (77)
Feeling cold (General disorders) | 4 (5)
Gait disturbance (General disorders) | 4 (4)
Influenza like illness (General disorders) | 3 (3)
Infusion site reaction (General disorders) | 1 (1)
Malaise (General disorders) | 6 (6)
Mucosal inflammation (General disorders) | 1 (1)
Nodule (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (5)
Oedema (General disorders) | 6 (7)
Oedema peripheral (General disorders) | 20 (24)
Pain (General disorders) | 5 (7)
Peripheral swelling (General disorders) | 1 (1)
Polyp (General disorders) | 1 (1)
Pyrexia (General disorders) | 28 (40)
Swelling (General disorders) | 1 (2)
Swelling face (General disorders) | 1 (2)
Systemic inflammatory response syndrome (General disorders) | 2 (3)
Thirst (General disorders) | 1 (1)
Ulcer (General disorders) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 3 (3)
Allergy to arthropod sting (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 3 (3)
Seasonal allergy (Immune system disorders) | 3 (3)
Acute sinusitis (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 9 (10)
Candida infection (Infections and infestations) | 8 (8)
Cellulitis (Infections and infestations) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3)
Cystitis (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 2 (2)
Fungal skin infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gingival abscess (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 6 (8)
Histoplasmosis (Infections and infestations) | 1 (1)
Histoplasmosis disseminated (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 4 (5)
Labyrinthitis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lymphangitis (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (2)
Nasal herpes (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 9 (12)
Nocardiosis (Infections and infestations) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 3 (3)
Oral herpes (Infections and infestations) | 4 (4)
Otitis externa (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 6 (7)
Pneumonia streptococcal (Infections and infestations) | 1 (1)
Pyuria (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2)
Rhinovirus infection (Infections and infestations) | 1 (1)
Root canal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 11 (13)
Skin infection (Infections and infestations) | 1 (3)
Soft tissue infection (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 26 (40)
Urinary tract infection (Infections and infestations) | 10 (13)
Viral infection (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (3)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 18 (23)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 10 (15)
Foreign body (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Muscle contusion (Injury, poisoning and procedural complications) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3)
Skin injury (Injury, poisoning and procedural complications) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 21 (54)
Amylase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 18 (29)
Blood alkaline phosphatase increased (Investigations) | 3 (4)
Blood bilirubin increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 7 (11)
Blood immunoglobulin g decreased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2)
Blood thyroid stimulating hormone increased (Investigations) | 3 (3)
Blood uric acid increased (Investigations) | 1 (1)
Heart rate irregular (Investigations) | 1 (1)
Immunoglobulins decreased (Investigations) | 2 (2)
Influenza a virus test positive (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (7)
Neutrophil count decreased (Investigations) | 4 (5)
Oxygen saturation decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 7 (11)
Protein total decreased (Investigations) | 1 (1)
Serum ferritin increased (Investigations) | 1 (1)
Tri-iodothyronine free decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 9 (11)
Weight increased (Investigations) | 2 (3)
White blood cell count decreased (Investigations) | 4 (6)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 42 (50)
Dehydration (Metabolism and nutrition disorders) | 13 (15)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 7 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (25)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (13)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (14)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (4)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (2)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 3 (3)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (25)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (25)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Groin pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (16)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 (10)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (11)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (11)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 (2)
Winged scapula (Musculoskeletal and connective tissue disorders) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 32 (37)
Dizziness postural (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (4)
Facial paralysis (Nervous system disorders) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 57 (71)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 10 (13)
Paraesthesia (Nervous system disorders) | 5 (5)
Parkinsonism (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 3 (3)
Sciatic nerve neuropathy (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 2 (3)
Sinus headache (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 4 (4)
Syncope (Nervous system disorders) | 2 (2)
Taste disorder (Nervous system disorders) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (4)
Alcoholism (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (6)
Confusional state (Psychiatric disorders) | 7 (7)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (4)
Dyssomnia (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 20 (21)
Mental status changes (Psychiatric disorders) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 5 (5)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 5 (5)
Haematuria (Renal and urinary disorders) | 6 (6)
Hypertonic bladder (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 3 (3)
Polyuria (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 3 (4)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Genital lesion (Reproductive system and breast disorders) | 1 (1)
Haematospermia (Reproductive system and breast disorders) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 44 (68)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (34)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 (15)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tracheal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (9)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (2)
Dandruff (Skin and subcutaneous tissue disorders) | 1 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (5)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (6)
Keloid scar (Skin and subcutaneous tissue disorders) | 1 (1)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 13 (14)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 7 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (15)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3)
Purpura (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 22 (37)
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 (6)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (10)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (3)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 5 (6)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1)
Skin sensitisation (Skin and subcutaneous tissue disorders) | 2 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (4)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 5 (5)
Hypertension (Vascular disorders) | 8 (10)
Hypotension (Vascular disorders) | 21 (23)
Lymphoedema (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Pallor (Vascular disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT02362035/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT02362035/SAP_001.pdf